CLINICAL TRIAL: NCT04683237
Title: Megestrol Acetate Versus Liraglutide Plus Megestrol Acetate in Obese Women with Endometrial Atypical Hyperplasia: a Randomized Controlled Pilot Clinical Study
Brief Title: Liraglutide Plus Megestrol Acetate in Endometrial Atypical Hyperplasia
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Based on our latest research results, we will revise the protocol and design a better study. Since no participants are enrolled till now, we withdraw this study.
Sponsor: Xiaojun Chen (Other)
Collaborators: Huashan Hospital (Other)
Responsible Party: Sponsor-Investigator, Xiaojun Chen, Principal Investigator, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 53211031
Record Dates: First submitted 2020-12-17; First posted 2020-12-24 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Atypical Endometrial Hyperplasia; Obese; Fertility Issues
MeSH Terms: conditions — Endometrial Hyperplasia; Obesity; Infertility | interventions — Liraglutide; Megestrol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MA alone (Other): enrolled patients will receive megestrol acetate 160mg po qd
  Interventions: Drug: Megestrol Acetate 160 MG
- MA+liraglutide (Experimental): enrolled patients will receive megestrol acetate 160mg po qd plus liraglutide (1.8mg/d or the max tolerable dosage)
  Interventions: Drug: Liraglutide Injection; Drug: Megestrol Acetate 160 MG

INTERVENTIONS:
Drug: Liraglutide Injection — Initiate liraglutide with a dose of 0.6 mg daily for one week. After one week at 0.6 mg per day, increase the dose to 1.2 mg daily in a week, and increase the dose to 1.8 mg daily after at least one week of treatment with the 1.2 mg daily dose. If the patients can not tolerate 1.8mg per day, decrease the dose to the max tolerable dose.
  Other Names: victoza; Nuo he li
  Arms: MA+liraglutide
Drug: Megestrol Acetate 160 MG — 160mg po qd
  Other Names: Yi li zhi; Megace

SUMMARY:
To investigate the efficacy of liraglutide plus megestrol acetate in obesity patients with atypical endometrial hyperplasia (AEH)

DETAILED DESCRIPTION:
Backgrounds: High-dose progesterone (MA/MPA) or LNG-IUS is the first-line treatment for women with atypical endometrial hyperplasia (AEH) or early endometrioid cancer who want to preserve fertility. About 70-80% of them can achieve complete response (CR) with the median time of 7-8 months. Over 10% of the patients can not achieve CR and choose operation finally. By the way, long-term treatment of progesterone has many side effects. Our previous study showed that overweight (BMI≥25kg/m2) AEH patients had a significantly increased risk of progesterone treatment failure, and the time to achieve CR is significantly prolonged. What's more, the greater the baseline weight of AEH patients, the greater the weight gains after high-dose progesterone treatment. Obese AEH patients have a lower response to high-dose progesterone. Weight management and lifestyle interventions are clearly written into 2020 uterine NCCN guidelines. We also find that metformin may improve insulin resistance in patients with AEH, and shorten time to achieve CR and increase the CR rates.

Liraglutide is a GLP-1 receptor agonist (GLP-1RA), which is one of the commonly used hypoglycemic drugs, has been approved for losing weight. And it is applicable for patients with BMI≥30 kg/m2 or ≥27 kg/m2 combined with one of the following: diabetes, hypertension, hyperlipidemia, sleep apnea. Liraglutide acts through improving insulin sensitivity, decreasing glucagon secretion , inhibiting appetite, delaying gastric emptying and improving whole-body inflammation condition.

Objective: To investigate whether liraglutide plus MA improve the efficacy of preserving fertility when compared to MA alone in obese women with AEH who want fertility conservation.

Design: A pilot prospective randomized controlled study is designed. And this study is open-label. We use SPSS (version 22.0,IBM) to design simple randomization. And participants will be randomly assigned (1:1) to receive MA alone or liraglutide plus MA. Patients in MA alone group will receive MA 160mg po qd and patients in the liraglutide plus MA group will receive liraglutide additionally with dose of 1.8mg/d or the max tolerance dose.

All enrolled patients will receive mentoring in weight management and lifestyle improvement. Hysteroscopic assessment will be performed every 12-16 weeks while other indexes will be evaluated every month, including weight, metabolic indications，inbody fat analysis, inflammation indicators and so on.

For the efficacy evaluation, CR is defined as the reversion of endometrial atypical hyperplasia to proliferative or secretory endometrium; partial response (PR) is defined as regression to simple or complex hyperplasia without atypia; no response (NR) is defined as the persistence of the disease; and progressive disease (PD) is defined as the appearance of endometrial cancer in patients. Continuous therapies will be needed in PR, NR or PD. Two months of maintenance treatment will be recommended for patients with CR, and participants will be followed up for 2 years.

Outcomes: Primary outcome is the CR rates of the two groups (MA alone VS MA+ liraglutide) . secondary outcomes include improvement of weight, insulin resistance, chronic inflammation condition, and time to achieve CR, and safety and side events during the therapy, and the recurrence rates, pregnancy rates and live birth rates in two years.

ELIGIBILITY:
Inclusion Criteria:

* BMI (body mass index) ≥28kg/m2
* Consent informed and signed
* Pathologically confirmed as endometrial atypical hyperplasia
* Have a strong desire to reproduce and ask for fertility preservation or those who insist on keeping the uterus despite no reproductive requirements
* Have good compliance and follow-up conditions, and patients are willing to follow up in Obstetrics and Gynecology Hospital of Fudan University in time

Exclusion Criteria:

* Diagnosed as type 2 diabetes
* Diabetic ketoacidosis
* History of acute pancreatitis
* Have a history or family history of medullary thyroid carcinoma; multiple endocrine neoplasia syndrome type 2 (MEN2)
* Combined with severe medical disease or severely impaired liver and kidney function
* Patients with other types of endometrial cancer or other malignant tumors of the reproductive system; patients with breast cancer or other hormone-dependent tumors that cannot be used with progesterone
* Those who require hysterectomy or other methods other than conservative treatment with drugs
* Deep vein thrombosis, stroke, myocardial infarction
* Smokers (≥15 cigarettes/day)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (CR) rates | From date of randomization until the date of CR, assessed up to 28 weeks.
  The 28-week CR rates will be calculated in two groups

SECONDARY OUTCOMES:
weight lose | From date of randomization until the date of CR, assessed up to 28 weeks
  weight changing in 28-week's intervention, weight will be recorded every 4 weeks.
changing of insulin resistance | From date of randomization until the date of CR, assessed up to 28 weeks.
  Glycated hemoglobin，Glucose tolerance test，Insulin release test，and C peptide release test will be performed at baseline and 28-week. During 12-16 week, fasting glucose, insulin, glycated hemoglobin and fasting C peptide will be tested once.
improvement of chronic inflammation | From date of randomization until the date of CR, assessed up to 28 weeks
  improvement of chronic inflammation indications in 28 weeks. In detail, indicators including TNF-α、IL-1, IL-6 and Creatine Kinase will be tested at 0,12-16th and 28th week.
Time of pathological complete response (CR) | From date of randomization until the date of CR, assessed up to 2 years.
  Time of histologic regression from AEH to proliferative or secretory endometrium
safety and side effects | From date of randomization until the date of CR, assessed up to 2 years.
  Adverse events related with Liraglutide and MA. Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 will be recorded, as well as incidence of adverse events.
Relapse rates | up to 2 years after the treatment for each patient
  All enrolled patients will be followed up for 2 years. During the following-up period, if patients recur after complete regression, they will be counted and the number of recurrence will be divided by number of patients followed up, then we can get the relapse rates.Comparison will be performed between two groups.
pregnancy outcomes | up to 2 years after the treatment for each patient
  For patients have a desire for fertility, pregnancies, births and related outcomes will be counted, and the rate of pregnancy will be counted as number of pregnancies/ number of patients trying to fertility in the following period. Comparison will be performed between two groups

CONTACTS AND LOCATIONS:
Overall Officials: xiaojun chen, Principal Investigator — Obstetrics & Gynecology Hospital of Fudan University

IPD SHARING:
Plan to Share IPD: No